CLINICAL TRIAL: NCT01736150
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Titration Study of Sevelamer Carbonate in CKD Patients on Hemodialysis
Brief Title: Dose-Titration Study of Sevelamer Carbonate in Chronic Kidney Disease (CKD) Patients on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVCARB03808
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease; Chronic Kidney Disease on Hemodialysis
Keywords: Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevelamer carbonate (Experimental): Subjects randomized by a central randomization system to one of two treatment groups in a 2:1 (active: placebo) fashion, stratified by Visit 1a phosphorus result (>5.5 mg/dL-6.5 mg/dL versus greater than 6.5 mg/dL), and site.
  Interventions: Drug: Sevelamer carbonate
- Placebo (Placebo Comparator): Subjects randomized by a central randomization system to one of two treatment groups in a 2:1 (active: placebo) fashion, stratified by Visit 1a phosphorus result (>5.5 mg/dL-6.5 mg/dL versus greater than 6.5 mg/dL), and site.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — * Starting dose of 1 tablet (800mg), three times per day (2.4g/day)with meals.
  * If serum phosphorus is higher than 5.5 mg/dL on Visit 3, 4, or 5, then dose increased by one additional tablet (800 mg). Three times daily with meals.
  Arms: Placebo
Drug: Sevelamer carbonate — * Starting dose 1 tablet (800 mg), three times per day (2.4 g/day) with meals.
  * If serum phosphorus is higher than 5.5 mg/dL on Visit 3, 4, or 5, then dose increased by one additional tablet(800mg).Three times daily with meals.
  Other Names: Renvela
  Arms: Sevelamer carbonate

SUMMARY:
The study aims to evaluate the efficacy and safety of sevelamer carbonate in reducing serum phosphorus and serum lipids (total and LDL-cholesterol) in Chronic Kidney Disease Patients on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* On hemodialysis regimen scheduled for four hour duration three times per week for a minimum 30 days prior to Visit 1 and throughout the study
* Have a central laboratory serum iPTH measurement less than 1000 pg/mL at Visit 1
* Have a central laboratory serum phosphorus measurement greater than 5.5 mg/dL at Visit 1a

Exclusion Criteria:

* Active dysphagia or swallowing disorder; or a predisposition to or current bowel obstruction, ileus, or severe gastrointestinal (GI) motility disorders including severe constipation
* Documented poorly controlled diabetes mellitus, poorly controlled hypertension, active vasculitis, human immunodeficiency virus infection, or any clinically significant unstable medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Visit 6/Early Termination (ET) in serum phosphorous. | 8 weeks
Frequency of treatment-emergent adverse events (AEs) and serious adverse events (SAEs), changes in laboratory parameters, and changes in vital signs. | 11 weeks

SECONDARY OUTCOMES:
Change from baseline to Visit 6/ET in serum lipids (total cholesterol and LDL-cholesterol). | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (18):
- China (18):
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital, Chengdu
  - Southwest Hospital, Chongqing
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Nanfang Hospital, Guangzhou
  - Sun Yat-Sen University School of Medicine 1st Affiliated Hospital, Guangzhou
  - Zhejiang University School of Medicine 1st Affiliated Hospital, Hangzhou
  - Jiangsu Province Hospital, Nanjing
  - Zhongda Hospital of Southeast University, Nanjing
  - Qingdao Municipal Hospital, Qingdao
  - Changzheng Hospital, Shanghai
  - Renji Hospital, Shanghai
  - Shanghai Ruijin Hospital, Shanghai
  - Xinhua Hospital, Shanghai
  - Zhongshan Hospital, Shanghai
  - Wenzhou College of Medicine 1st Affiliated Hospital, Wenzhou